CLINICAL TRIAL: NCT05794555
Title: LiveSMART: A Sequential, Multiple Assignment Randomized Trial to Prevent Falls in Patients With Cirrhosis
Brief Title: LiveSMART Trial to Prevent Falls in Patients With Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Elliot B. Tapper, Associate Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HUM00225275; CER-2021C3-24907 (Other: PCORI)
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cirrhosis, Liver; Portal Hypertension
Keywords: Exercise program; Lactulose; Tai-Chi; Fall prevention; Dietary Protein
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Lactulose

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in stage 1 to enhanced usual care or enhanced usual care plus lactulose. After 12 weeks participants will be re-randomized to TeleTai-Chi (at-home, via Zoom, supervised by a study team instructor) vs. continued enhanced usual care. The participants that took lactulose in Stage 1 will continue to take lactulose through Stage 2 until their participation is complete. The caregivers (of the trial participants) involved in the observational sub-study are not included in the trial in any fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Enhanced Usual Care group followed by investigator recommended exercise (Active Comparator): Enhanced Usual Care (EUC) at Stage 1 (12 weeks) and then re-randomization to EUC then Investigator-Recommended Exercise at Stage 2
  Interventions: Behavioral: Enhanced Usual Care; Behavioral: Investigator recommended exercise
- Treatment (Lactulose) plus Enhanced Usual Care then TeleTai-Chi exercise classes (Experimental): Lactulose plus Enhanced Usual Care (EUC) at Stage 1 (12 weeks) and then re-randomization to Lactulose plus EUC then TeleTai-Chi exercise classes at Stage 2
  Interventions: Behavioral: Enhanced Usual Care; Drug: Lactulose; Behavioral: TeleTai-Chi (virtual)
- Enhanced Usual Care group followed by Tele-Tai Chi exercise classes (Experimental): Enhanced Usual Care (EUC) at Stage 1 (12 weeks) and then re-randomization to EUC then Tele-Tai Chi exercise classes at Stage 2
  Interventions: Behavioral: Enhanced Usual Care; Behavioral: TeleTai-Chi (virtual)
- Treatment (Lactulose) plus Enhanced Usual Care then recommended exercise (Experimental): Lactulose plus Enhanced Usual Care (EUC) at Stage 1 (12 weeks) and then re-randomization to Lactulose plus EUC then Investigator-Recommended Exercise at Stage 2
  Interventions: Behavioral: Enhanced Usual Care; Drug: Lactulose; Behavioral: Investigator recommended exercise

INTERVENTIONS:
Behavioral: Enhanced Usual Care — Patients will be provided and counseled on two methods which will enhance care. The first is a handout on nutrition recommendations and protein supplementation. This will include the recommendation of both high protein snacks during the daytime (e.g., protein bars) and a high-protein night-time snack (e.g., peanut butter and crackers). The second will be to counsel participants on falls prevention methods that can be enacted in day-to-day life. All participants will be provided with a standard hand-out of Centers for Disease Control and Prevention (CDC)-endorsed fall-risk reduction measures.
Drug: Lactulose — Patients will be prescribed lactulose and will also receive enhanced usual care. Lactulose will be taken on a specific schedule based on the average number of bowel movements on average per day. It will be started at 15 milliliter (mL) dose and will be instructed to slowly increase the lactulose dose over the course of the first week of Stage 1 participation. The prescribed maximum dose will be 30 mL (20g) twice daily. The dose will slowly increase toward the maximum or until participants reach 2-3 soft bowel movements daily.
  Participants that receive Lactulose during stage 1 will continue this in stage 2.
  Arms: Treatment (Lactulose) plus Enhanced Usual Care then TeleTai-Chi exercise classes; Treatment (Lactulose) plus Enhanced Usual Care then recommended exercise
Behavioral: Investigator recommended exercise — Participants randomized to enhanced usual care will be reminded of standard fall precautions outlined in the Fall Prevention Primer that were provided in Stage 1 and will receive exercise recommendations.
  Arms: Enhanced Usual Care group followed by investigator recommended exercise; Treatment (Lactulose) plus Enhanced Usual Care then recommended exercise
Behavioral: TeleTai-Chi (virtual) — TeleTai-Chi will be taught remotely via live Zoom classes of up to 15 patients by a certified TeleTai-Chi instructor three times per week (for approximately 12 weeks). Classes will be conducted via a HIPAA-compliant Zoom server through the University of Michigan. Participants will be instructed to use Zoom by smartphone, tablet, or computer. High-Definition Multimedia Interface (HDMI) cables and other device specific equipment to connect devices to televisions will be provided.
  Arms: Enhanced Usual Care group followed by Tele-Tai Chi exercise classes; Treatment (Lactulose) plus Enhanced Usual Care then TeleTai-Chi exercise classes

SUMMARY:
This multicenter trial is being conducted to determine if sequential lactulose and Tele (virtual) Tai-Chi reduces the rate of injurious fall, non-injurious falls, incident overt Hepatic Encephalopathy (HE), and death or liver transplant over 24 weeks.

Participants that are enrolled will be randomized to stage one of this project for approximately 12 weeks. After completing stage one, participants will be re-randomized to stage 2 of the project that will last approximately 12 more weeks.

The study hypothesizes that sequential lactulose/TeleTai-Chi will reduce falls, incident overt HE, death and physical frailty and will improve cognitive function, and Health Related Quality of Life (HRQOL) over 24 weeks compared to other treatment combinations.

As detailed below, an observational component that enrolls caregivers of the trial participants is being conducted. Upon completion, Participants listed in the record here only include trial participants; and the observational component was moved to a new registration for clarity, NCT07140120.

DETAILED DESCRIPTION:
The Clinicaltrials.gov registration record was updated as requested by Patient-Centered Outcomes Research Institute (PCORI) based on protocol amendment version 3.0 after approval by the Institutional Review Board. These changes included: the additional aim for a supplemental observational study to assess social determinants of health, financial burdens, etc., and includes recruitment of the caregivers for this supplemental study along with the trial participants, as well as updated outcomes for the trial. After further discussion with PCORI, these changes were removed from this record and used to create a separate record for the supplemental study focused on caregivers (NCT07140120).

The caregivers that are enrolled are not in the clinical trial. All clinical trial information is provided in this record, but upon completion of enrollment and consideration of transparent results reporting, it was decided to move all the items related to the observational supplemental study to its own record.

To improve clarity in the record, the two arms representing stage 1 of the project were incorporated into the remaining four representing stage 2, so the remaining arms now represent both stage 1 and stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cirrhosis based on histology and/or imaging specified in the protocol.
* Evidence of portal hypertension - must meet at least one of the following criteria:

  * Ascites (present or within past 2 years)
  * Varices (seen by Esophagogastroduodenoscopy or by Ultrasound(US) or cross-sectional imaging)
  * Fibroscan Liver stiffness measurement (LSM) >25 kilopascals (kPa) (if no other factors present)
  * Magnetic resonance elastography (MRE) LSM > 5 kPa (if no other factors present)
  * Acoustic radiation force impulse LSM > 17kpa (if no other factors present)
  * Hepatic vein pressure gradient > 10 millimetres of mercury (mmHg)
  * Portal hypertensive gastropathy seen on Esophagogastroduodenoscopy
  * Platelet count < 80/ units per liter (uL)
  * Recanalized umbilical vein (by US or cross-sectional imaging)
* Access to Wireless Fidelity (Wi-Fi) at home
* Owns or access to a smartphone, tablet or computer
* English or Spanish speaking
* Willing to participate in exercise program

Exclusion Criteria:

* Overt hepatic encephalopathy (HE) within 6 months, requiring >28 days total of lactulose
* Took lactulose for non - HE reasons for >28 days total in last 6 months
* Took Rifaximin for > 28 days total in last 6 months
* Model for End Stage Liver Disease (MELD) > 25 (Exception: MELD > 25 with clinically stable End-Stage Renal Disease (ESRD) for whom the bilirubin is < 5 g/dL)
* Barcelona Clinic Liver Cancer (BCLC) > C Hepatocellular Carcinoma (HCC)
* Currently taking Sorafenib, Atezolizumab/Bevacizumab, Regorafinib, or Cabozatinib
* Greater than (>) 3 paracentesis/month in last 2 months
* Active Metastatic solid malignancy or acute leukemia within last 3 years
* Severe cognitive, vision, or hearing impairment (without use of corrective lenses or hearing assist devices) or psychiatric illness precluding study participation
* Currently participates in Tai-Chi or performs >150 min/week vigorous physical activity
* Currently receiving lower body physical and/or occupational therapy
* Living in an assisted living facility
* Hemoglobin A1C > 12 (within past 12 months)
* Requires a low galactose diet
* Deemed unsuitable by the study investigator

Inclusion Criteria for the Caregivers of the participants:

* Adult > 18 years of age
* Informal caregiver of a participant enrolled in LIVE-SMART
* English speaking

Exclusion Criteria for the Caregivers of the participants:

- Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing a hierarchical composite of events over 24 weeks: injurious falls, non-injurious falls, incident Hepatic Encephalopathy, liver transplant, and death/transplant | Baseline to 24 weeks (following stage 2)
  Composite outcome is defined as any of the following:
  • Injurious Fall: Fracture, dislocation, cut, head injury, soft - tissue injury requiring medical intervention including: Hospitalization or overnight observation in the Emergency Room (ER); surgery, transfusion, stitches
  * Non - Injurious Fall: Inadvertently coming to rest on the floor or lower level
    * Include falls that result in minor injuries that are addressed with first aid (e.g., ice, bandage)
  * Incident Overt HE: Acute disorientation requiring hospitalization or the initiation of HE - directed therapy, confirmed by a gastroenterologist or study investigator
  * Death: Mortality with any cause
  * Liver transplant: Replacement of a diseased liver with the healthy liver from another person because of acute-on-chronic liver failure (using the EASL-CLIF-C definition consisting of an acute increase in the bilirubin and/or INR, acute kidney injury, overt HE, hypertension, and hypoxia).

SECONDARY OUTCOMES:
Injurious Falls | Baseline to 24 weeks (following stage 2)
  Falls include: Fracture, dislocation, cut, head injury, soft - tissue injury requiring hospitalization.
Non-Injurious Falls | Baseline to 24 weeks (following stage 2)
  Non- Injurious Falls include: Inadvertently coming to rest on the floor or lower level
Incident Overt hepatic encephalopathy (HE) | Baseline to 24 weeks (following stage 2)
  Incident Overt HE includes: Acute disorientation requiring hospitalization or the initiation of HE - directed therapy, confirmed by a gastroenterologist or study investigator.
Death/transplant | Baseline to 24 weeks (following stage 2)
  Mortality with any cause or liver transplantation
Incident of Liver Transplant | Baseline to 24 weeks (following stage 2)
  Replacement of a diseased liver with the healthy liver from another person.
Days-alive and out-of-the-hospital | Baseline to 24 weeks (following stage 2)
  Days-alive and out-of-the-hospital is a continuous value, 1 for each day alive, 0 for days in hospital. Participants will be queried and data will also be abstracted from the Electronic Medical Record (EMR).
Cognitive Function based on the Animal Naming Test (ANT) | Baseline to 24 weeks (following stage 2)
  The animal naming test assesses cognitive function. It is a timed test that that consists of participants listing as many unique animals as possible in 60 seconds. This is a validated test used for the assessment of hepatic encephalopathy. The score is the number of unique animals stated (higher is better).
Visual Analog Scale (VAS) | Baseline to 24 weeks (following stage 2)
  This is a 1-item global rating of health scored 0-100. A score of 100 means the best health and 0 means the worst health imagined.
The Patient Reported Outcome Measurement Information System (PROMIS)-29+2 v2.1 | Baseline to 24 weeks (following stage 2)
  There are seven health domains including physical function, anxiety, depression, fatigue, sleep disturbances, ability to participate in social roles and activities, and pain interference. Each category consists of 4 questions. Questions are ranked on a 5-point Likert scale, with higher scores at times indicating better quality of life, and at other times indicating poorer quality of life. There is a pain rating scale ranging from 0 to 10, with higher scores indicating higher pain level.
Depression based on The Patient Reported Outcome Measurement Information System (PROMIS)-29+2 v2.1 | Baseline to 24 weeks (following stage 2)
  There are 4 questions that participants complete regarding depression (never 1 - always 5). Scoring ranges (4-20) with higher scores indicating more depression.
Sleep quality based on the PROMIS-29+2 v2.1 | Baseline to 24 weeks (following stage 2)
  There are 4 questions and are ranked on a 5-point Likert scale (not at all or very poor 1 - 5 very much). Scoring ranges (4-20) with lower scores indicating better sleep quality.
Physical frailty based on the Liver Frailty Index | Baseline to 24 weeks (following stage 2)
  Physical frailty will be assessed with this index and is a composite of handgrip, timed chair-stands, and balance. The index ranges from -1.26 (robust) to 6.9 (frail), 50th percentile is 3.9. For individuals enrolled remotely, the study team will assess chair-stands.
Physical frailty based on the Activities of daily living (ADLs) | Baseline to 24 weeks (following stage 2)
  Activities of daily living (ADLs), is a validated self-reported measure (disability is defined as >1 ADL deficit) recommended by the American Society for Transplantation and AASLD
Intervention Fidelity | 12 and 24 weeks
  Evaluation of intervention fidelity will be assessed at 50% and 100% of study completion as percent delivery of key intervention components including coordinator trainings, lactulose prescriptions ordered, enhanced usual care components delivered, Short Message Service (SMS) assessments sent, study visits completed, and exercise sessions completed.
Participant adherence | 12 weeks and 24 weeks
  Adherence to lactulose, Tai-Chi, and nighttime protein supplementation will be monitored. Adherence is the proportion of expected-to-actual treatment days completed during the intervention.
Participant satisfaction with the trial and interventions based on the Patient Global Impression of Change (PGIC) | 12 weeks and 24 weeks
  Satisfaction with the trial will be assessed using the 6-item Patient Global Impression of Change (PGIC). Participants select from Very much improved 1 - Very much worse 7. Lower scores indicate higher satisfaction.
Short Form (SF) - 8 | 12 weeks and 24 weeks
  The SF-8 is an abbreviated 8-item version of an original 36-item health survey (SF-36). It is a generic multipurpose quality of life instrument. It contains psychometrically based physical and mental health summary measures. The eight domains include general health, physical functioning, role physical, bodily pain, vitality, social functioning, mental health and role emotional. The scores range 8-40, with a lower score meaning higher function.

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Tapper, MD, Principal Investigator — University of Michigan; Marina Serper, MD, MS, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Scott & White Research Institute (BSW), Dallas, Texas